CLINICAL TRIAL: NCT01513564
Title: Multimodal Perioperative Pain Management of Circumferential Lumbar Fusion Improves Recovery
Brief Title: Multimodal Perioperative Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Vejle Hospital (Other); Aarhus University Hospital (Other); Copenhagen University Hospital, Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: ON-07-008-RAS
Record Dates: First submitted 2011-12-13; First posted 2012-01-20 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Degenerative Spondylolisthesis
Keywords: Disc disease; Spondylolisthesis
MeSH Terms: conditions — Spondylolisthesis | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Conservative treatment program (Experimental): The control group were supervised isometric passive and active exercises by a physiotherapist. On the second day patients were allowed to sit in a chair being instructed to a low intensity exercise training program with regard to back pain and fear of activity. From the third or fourth day stair training, low intensity exercise, daily walks and instruction in home training were allowed.
  The intervention group received the same training program but with a faster program plus a higher intensity exercise-training program.
  Interventions: Drug: Postoperative epidural morphine; Drug: Local anaesthesia

INTERVENTIONS:
Drug: Postoperative epidural morphine — The control group received postoperative epidural morphine 0.4 mg/ml four times a day, epidural bupivacaine 2.5 mg/ml, 3-4 ml on request for 75 hours and a 7 day rehabilitation program.
  Other Names: Convalescence after lumbar fusion
Drug: Local anaesthesia — Preemptively and posteruptively, the intervention group received local anaesthesia with bupivacaine 2.5 mg/ml, 10 + 10 ml posteriorly and 10 + 10 anteriorly; preemptive epidural analgesia with 3 ml lidocaine 20 mg/ml, 3 ml, 10 ml morphine 0.4 mg/ml plus 5 ml bupivacaine; postoperative continuous epidural analgesia for 72 hours with 250 ml with bupivacaine 1 mg/ml + morphine 50 ug/ml, and 0.5 ml epinephrine 1 mg/ml, 4 ml/hour, and after wound closure ketorolac 30 mg intravenously.
  Other Names: Convalescence after lumbar fusion.

SUMMARY:
Convalescence after lumbar fusion is dependent on pain. In orthopaedic and abdominal surgery accelerated stay programs with optimized pain management enhance recovery.

The objective is to evaluate the effect of a revised and optimized perioperative fast track program in lumbar fusion surgery.

DETAILED DESCRIPTION:
Major spine surgery is usually associated with high postoperative pain scores and opioid requirements. Epidural analgesia has been reported to be an effective and safe method to control postoperative pain after spinal instrumentation surgery, but the overall effects of pain management on postoperative length of stay and recovery remains debatable.

However, in a multimodal approach, including multimodal non-opioid analgesia to control postoperative pathophysiology and rehabilitation, complications and hospital stay have been reduced after arthroscopy, hip arthroplasty and knee arthroplasty, hip fractures and abdominal surgery and other procedures, when combined with an enhanced recovery program.

The aim of the study is to assess the effect and safety of a combined analgesic regimen consisting of local anesthetic, intra-operative and post-operative continuous epidural analgesia and a single dose ketorolac together with a fast track rehabilitation program after 360 degree lumbar fusion for degenerative disc disease and spondylolisthesis < 2

ELIGIBILITY:
Inclusion Criteria:

* Degenerative disc disease and Spondylolisthesis up to grade 2 at one to the three lower lumbar levels.

Exclusion Criteria:

* Previous fusion, metabolic bone disease, severe comorbidity or psychological instability.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-01; Primary Completion 2003-12 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Multimodal management of lumbar fusion | Two years
  Back and leg pain on VAS, neurological deficits, hospital stay, bony fusion and Oswestry Disability Index

SECONDARY OUTCOMES:
Multimodal management of lumbar fusion | Two years
  Assessment of the effects of at fast track program with ongoing epidural analgesia, multimodal pain treatment including ketorolac and early intensive mobilization and physiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D., Principal Investigator — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark; David S. Krum-Moeller, M.D., Study Chair — Department of Orthopaedic Surgery, Vejle and Give Hospital; Lene R. Lauridsen, Study Chair — Department of Orthopaedic Surgery, Vejle and Give Hospital; Henrik Kehlet, M.D., Study Chair — Section for Surgical Pathophysiology, Juliane Marie Centre, Rigshospitalet, Copenhagen
Locations (1):
- Orthopaedic Research Unit, Aarhus University, Aalborg Hospital, Aalborg, Denmark